CLINICAL TRIAL: NCT04651673
Title: Behandlingseffekter Med Avlastande knäortoser för Patienter Med knäartros En Retro-och Prospektiv Multicenterregisterstudie
Brief Title: Prescribed Knee Brace Treatments for Osteoarthritis of the Knee (Knee OA)
Status: Enrolling by invitation | Type: Observational
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: CIP2020050839
Record Dates: First submitted 2020-11-18; First posted 2020-12-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee brace; conservative treatment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: This is a non interventional registry — All patients, at listed investigational sites, that get prescription for a knee orthosis indicated for Knee OA symptomatic treatment, get an invite to partake in the evaluation registry.

SUMMARY:
The study is a non-controlled retro- and prospective multi center patient registry study.

Subjects will be given a study ID number assigned at first brace fitting after consenting to partake. Participants will be asked to fill in a questionnaire either in electronic or paper version at first fitting. Additional follow up questionnaires will be implemented at 4 weeks, 6 months and 1 year post initial brace fitting. After that period patients will be contacted every year, until brace termination/ knee surgery or death.

DETAILED DESCRIPTION:
This is a noninterventional registry study pertaining to knee OA braces. There are no comparative devices or treatments. Subjects are expected to follow the recommendations of the brace subscriber and other health care professionals at any time independent of their continuation within the registry.

Subjects will be enrolled at the clinic where their brace was prescribed or at the site where the brace was fitted.

There is no formal end date for this data registry. A revisit to this protocol may be motivated after 5 years, to assess if longer follow up is required.

For individual participants follow up will continue with annual questionnaires as long as the brace is in use. The questionnaires will be administered either through mail with a paper version, or through a link to an electronical version (ePRO). There is also a possibility of administrating the questionnaires as a phone guided interview, if that is a mean that serves the patient or clinics better. The planned follow-ups are at 4 weeks, 6 months, 1 year from brace prescription and then annually as long as participants are disposed as "ongoing" in the registry.

The questionnaires contains question about pain, function, medication, general brace use and quality of life question.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are prescribed knee brace for symptomatic treatment of knee OA from partaking clinics
* Older than 18 years

Exclusion Criteria:

* Younger than 18 years
* Not willing or able to sign informed consent, or not cognitive impairments preventing understanding of the questionnaires.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are patients that have been prescribed knee braces for treatment of knee OA. The brace prescription is independent of the registry, i.e. no one is prescribed a brace because of the registry or for the purpose of this data collection per se
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that are using the braces | 6 months follow up
  brace usage, days per week
Change in Pain status compared to baseline | 6 months follow up
  Knee injury and Osteoarthritis Outcome Score (KOOS)-12
Change in Mobility compared to baseline | 6 months follow up
  KOOS-12
Proportion of patients that are still using the braces | 1 year follow up
  brace usage, days per week
Change in Pain status compared to baseline | 1 year follow up
  KOOS-12
Change in Mobility compared to baseline | 1 year follow up
  KOOS-12
Sick leave after receiving the braces | 6 months follow up
  Proportion of sick leave
Sick leave after receiving the braces | 1 year follow up
  Proportion of sick leave
Changes in reported quality of life | 6 months follow up
  KOOS-12
Changes in reported quality of life | 1 year follow up
  KOOS-12
Changes in QALY's | 6 months follow up
  EQ-5D-5L
Changes in QALY's | 1 year follow up
  EQ-5D-5L

OTHER OUTCOMES:
The patients' satisfaction of the value/effectiveness of the brace | 6 months follow up
  Numeric Rating Scale (NRS) for satisfaction (0-10)
The patients' satisfaction of the value/effectiveness of the brace | 1 year follow up
  NRS for satisfaction (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Dencker, Dr, Principal Investigator — Region Skåne
Locations (1):
- Skånevård Nordost Region Skåne - Verksamhets område ortopedi, Kristianstad /Hässleholm, Hässleholm, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No